CLINICAL TRIAL: NCT01511978
Title: Inpatient Double-Blind Placebo-Controlled Withdrawal Study of 3,4-Diaminopyridine Base (3,4-DAP) in Subjects With Known Lambert-Eaton Myasthenic Syndrome
Brief Title: Effectiveness of 3,4-Diaminopyridine in Lambert-Eaton Myasthenic Syndrome
Acronym: DAPPER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jacobus Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JPC 3,4-DAPPER
Record Dates: First submitted 2011-12-24; First posted 2012-01-19 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Lambert-Eaton Myasthenic Syndrome; Eaton-Lambert Myasthenic Syndrome
Keywords: Lambert-Eaton; Eaton-Lambert; myasthenia; myasthenic; LEMS; LES; DAP; diaminopyridine; 3,4-diaminopyridine; 3,4-DAP
MeSH Terms: conditions — Lambert-Eaton Myasthenic Syndrome | interventions — Amifampridine

STUDY DESIGN:
Intervention Model Description: This was a multicenter, randomized, double-blind, placebo-controlled withdrawal study to assess the safety and efficacy of 3,4-DAP in subjects on a stable regimen of all LEMS-related treatments, including 3,4-DAP, for a minimum of 3 months prior to study entry. Subjects who met all study entry criteria were randomized in a 1:1 ratio to continue their current treatment regimen (Group A, continuous 3,4-DAP) or tapered withdrawal from 3,4-DAP (Group B, taper to placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Continuous 3,4-DAP (Active Comparator): Subjects continued taking their usual individualized regimen of 3,4-DAP base, 30 to 100 mg daily divided into at least 3 doses.
  Interventions: Drug: Continuous 3,4-DAP
- Taper 3,4-DAP to Placebo (Placebo Comparator): Subjects were tapered over 3 days from their usual individualized regimen of 3,4-DAP base (30 to 100 mg daily divided into at least 3 doses) to placebo with up to an additional 16 hours of placebo before resuming their usual pre-study regimen of 3,4-DAP base
  Interventions: Drug: Taper 3,4-DAP to Placebo

INTERVENTIONS:
Drug: Continuous 3,4-DAP — Subjects were maintained on their usual personal dose and schedule of 3,4-DAP base
  Other Names: 3,4-Diaminopyridine; 3,4-Pyridinediamine; Diamino-3,4-pyridine
  Arms: Continuous 3,4-DAP
Drug: Taper 3,4-DAP to Placebo — Subjects were tapered over 3 days from their usual regimen of 3,4-DAP base to placebo with up to an additional 16 hours of placebo before resuming their usual pre-study regimen of 3,4-DAP base
  Other Names: 3,4-Diaminopyridine; 3,4-Pyridinediamine; Diamino-3,4-pyridine; Placebo
  Arms: Taper 3,4-DAP to Placebo

SUMMARY:
Hypothesis: 3,4-Diaminopyridine base (3,4-DAP) improves Lambert-Eaton Myasthenic Syndrome (LEMS)-related weakness.

DETAILED DESCRIPTION:
The objectives of the study were to confirm the safety and to test the efficacy of 3,4-DAP in the treatment of LEMS-related weakness.

This was a phase 2 randomized double-blind placebo-controlled withdrawal study in subjects with known clinically active LEMS who had been on a chronic stable dose of compassionate distribution Jacobus 3,4-DAP provided through FDA-approved individual investigator-held INDs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or over
2. Ambulatory while taking 3,4-DAP, i.e. the patient was able to perform the timed up and go (TUG), either with or without an assistive device
3. Established diagnosis of LEMS, with documentation provided
4. Continuous use of Jacobus 3,4-DAP for at least 3 months
5. Minimum of 3 doses per day with no single dose less than 10 mg of 3,4-DAP
6. The patient needed to wait about 15 to 30 minutes to experience an unequivocal improvement in a LEMS-induced dysfunction after they take their first dose of 3,4-DAP in the morning [a patient who remains in bed past this point by choice may still be eligible]
7. Stable regimen of all LEMS-related treatments for at least 3 months
8. Stable daily regimen of other medications (prescription and over-the-counter) for a minimum of 1 month
9. Willing to chance being tapered off of 3,4-DAP
10. Fluency in English
11. If applicable, agreed to use birth control during heterosexual intercourse until at least 2 weeks after completion of study
12. A signed informed consent by the study subject

Exclusion Criteria:

1. Last monoclonal antibody treatment (e.g. rituximab) was less than 6 months ago (i.e., recent treatment is an exclusion)
2. Clinically significant or poorly controlled condition that in the opinion of the study personnel might pose an unacceptable risk to the patient if entered into the study
3. Respiratory failure requiring intubation while on 3,4-DAP with no precipitating event or medication
4. Use of any investigational drug other than 3,4-DAP within the last 30 days
5. Pregnant or lactating
6. Current use of other aminopyridines (e.g.4-AP) or guanidine
7. Did not display a sufficiently large response to 3,4-DAP during the baseline observation period in the CRU to detect a decline during withdrawal of 3,4-DAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy L Aleš, MD, Study Director — Jacobus Pharmaceutical
Locations (7):
- United States (7):
  - University of California at Davis, Sacramento, California
  - Indiana University, Indianapolis, Indiana
  - Duke University, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were referred by active Investigational New Drug (IND) holders involved with the Jacobus Pharmaceutical Company's 3,4-diaminopyridine (3,4-DAP) free base compassionate distribution program.
Pre-assignment Details: 52 patients were assessed for eligibility. 20 were ineligible. 32 were randomized and completed the study.
Groups:
- Continuous 3,4-DAP: Subjects were administered their usual dosage on their regular personalized schedule
- Taper 3,4-DAP to Placebo: Subjects were administered decreasing amounts of 3,4-DAP on their regular personalized schedule
Period: Overall Study
Arm/Group | Continuous 3,4-DAP | Taper 3,4-DAP to Placebo
Started | 14 | 18
Completed | 14 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Continuous 3,4-Diaminopyridine (3,4-DAP): Subjects were administered their usual dosage on their regular personalized schedule
- 3,4-DAP Taper to Placebo: Subjects were administered decreasing amounts of 3,4-DAP on their regular personalized schedule
- Total: Total of all reporting groups
Arm/Group | Continuous 3,4-Diaminopyridine (3,4-DAP) | 3,4-DAP Taper to Placebo | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (15.97) | 59.3 (14.99) | 55.5 (15.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 17 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 11 | 18 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 168.5 (5.67) | 169.6 (8.98) | 169.2 (7.67)
Weight [Mean (Standard Deviation); unit: kg] | 78.0 (19.11) | 80.3 (18.95) | 79.3 (18.73)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.3 (5.92) | 27.7 (5.14) | 27.5 (5.39)
Age at diagnosis [Mean (Standard Deviation); unit: years] | 44.1 (13.79) | 52.7 (14.76) | 48.9 (14.76)
Time between symptom onset and diagnosis [Mean (Standard Deviation); unit: years] | 0.9 (0.62) | 2.2 (3.00) | 1.7 (2.35)
Duration of diagnosis prior to randomization [Mean (Standard Deviation); unit: years] | 6.7 (5.70) | 6.7 (6.08) | 6.7 (5.82)
Positive P/Q type voltage-gated calcium channel (VGCC) antibodies at screening [Count of Participants; unit: Participants] | 12 | 17 | 29
Compound Muscle Action Potential (CMAP) consistent with Lambert-Eaton Myasthenia (LEM) at screening [Count of Participants; unit: Participants] | 7 | 10 | 17
Total Daily Dose of 3,4-DAP at randomization [Median (Full Range); unit: mg] | 80.0 [35 to 100] | 80.0 [30 to 100] | 80 [30 to 100]
Number of 3,4-DAP individual daily doses at randomization [Median (Full Range); unit: number of daily doses] | 4.5 [3 to 7] | 5.0 [3 to 6] | 5.0 [3 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 30% or More Deterioration in Triple Timed Up & Go (3TUG) Test, Compared to Time-matched Baseline
Description: The 3TUG time obtained 2 hours after the last dose of the withdrawal period (i.e., at time of theoretical "peak drug effect") was compared to the average time-matched 3TUG tests performed during 2 days of baseline observation prior to randomization.
  The study endpoint was a change of more than 30% in the final post-dose 3TUG during the withdrawal period and was based on blinded readings of video recordings of 3TUG tests.
Time Frame: Baseline period (days 0, 1, 2); Randomized treatment period (starting with last dose of day 2, and days 3, 4, 5, and ending with first dose on day 6 when pre-randomization regimen was resumed, or rescue, if indicated sooner)
Measure: Count of Participants; unit: Participants
Groups:
- Continuous 3,4-Diaminopyridine (3,4-DAP): Subjects were continued on their usual pre-randomization 3,4-DAP dosing regimen.
- 3,4-DAP Taper to Placebo: Subjects were tapered off of their pre-randomization 3,4-DAP dosing regimen over 3 days with up to an additional 16 hours of placebo.
Arm/Group | Continuous 3,4-Diaminopyridine (3,4-DAP) | 3,4-DAP Taper to Placebo
Number analyzed (Participants) | 14 | 18
Participants | 0 | 13
Statistical Analysis 1: Comparison: Continuous 3,4-Diaminopyridine (3,4-DAP) vs 3,4-DAP Taper to Placebo; Test type: Superiority; p < 0.0001, Fisher Exact

2. Secondary Outcome: Self-assessment of LEMS-related Weakness, W-SAS
Description: The last post-dose self-assessment of LEMS-related weakness from the withdrawal period with categories of much much weaker (-3), much weaker (-2), somewhat weaker (-1), about the same (0), somewhat stronger (1), much stronger (2), and much much stronger (3).
Time Frame: Participants were followed for up to 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 3,4-DAP: Subjects were administered their usual dosage on their regular personalized schedule.
Arm/Group | 3,4-DAP | 3,4-DAP Taper to Placebo
Number analyzed (Participants) | 14 | 18
units on a scale | -0.2 (1.24) | -2.4 (0.85)
Statistical Analysis 1: Comparison: 3,4-DAP vs 3,4-DAP Taper to Placebo; Test type: Superiority; p = 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the inpatient stay of up to 7 days on the clinical research unit and then weekly with standard telephone follow-up and diary entries for one month following discharge from the clinical research unit.
Description: The return of Lambert-Eaton Myasthenic Syndrome (LEMS)-related signs and symptoms in a withdrawal design was anticipated and therefore adverse events were categorized as (1) treatment emergent adverse events, (2) treatment emergent adverse events excluding LEMS-related signs and symptoms, and (3) LEMS-related signs and symptoms adverse events
Arm/Group | Continuous 3,4-Diaminopyridine (3,4-DAP) | 3,4-DAP Taper to Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/18
Other Adverse Events (participants affected / at risk) | 5/14 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous 3,4-Diaminopyridine (3,4-DAP) (N=14) | 3,4-DAP Taper to Placebo (N=18)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Hospitalization for pneumonia occurred one month following discharge from the clinical research unit and was consider not related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continuous 3,4-Diaminopyridine (3,4-DAP) (N=14) | 3,4-DAP Taper to Placebo (N=18)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Sjogren (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Injection site bruising (General disorders) | 1 | 0
Instillation site irritation (General disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication shall be a multicenter publication submitted after conclusion of the Study at all sites. If a multicenter publication is not submitted within 12 months, PIs may use results.

The only other disclosure restriction on the PI is that the Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of 30 days for confidential review. This period may be extended by 60 days at Sponsor's request.